CLINICAL TRIAL: NCT00592306
Title: A Prospective Single Center Randomized Trial of Intraoperative Versus Postoperative Thymoglobulin in Lung Transplantation.
Brief Title: Intraoperative Versus Postoperative Thymoglobulin in Lung Transplantation
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: University of California, Los Angeles (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ATG in Lung Transplantation
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Lung Transplant
Keywords: ATG; rabbit thymoglobulin; reperfusion lung injury; primary graft dysfunction; lung transplantation
MeSH Terms: conditions — Primary Graft Dysfunction | interventions — thymoglobulin; Postoperative Period

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- thymoglobulin (intraoperative) (Active Comparator): we plan to blindly randomize these 25 lung transplant patients to intraoperative dosing of thymoglobulin followed by 3 additional postoperative doses (the first of these 3 postoperative doses will be placebo)
  Interventions: Drug: thymoglobulin (intraoperative)
- thymoglobulin (postoperative dosing) (Placebo Comparator): We plan to blindly randomize these 25 lung transplant patients to 3 postoperative doses of thymoglobulin (the intraoperative dose will be placebo)
  Interventions: Drug: thymoglobulin (postoperative)

INTERVENTIONS:
Drug: thymoglobulin (intraoperative) — All patients (Arm I and Arm II) will receive 3 doses of thymoglobulin at 1.5mg/kg IV over 6 hours; only the timing of the medication is being altered.
  Each arm will also receive a single placebo dose.
  Arm I will receive thymoglobulin intraoperatively followed by a postoperative placebo dose and two subsequent thymoglobulin doses.
  Other Names: thymoglobulin
  Arms: thymoglobulin (intraoperative)
Drug: thymoglobulin (postoperative) — All patients (Arm I and Arm II) will receive 3 doses of thymoglobulin at 1.5mg/kg IV over 6 hours; only the timing of the medication is being altered.
  Each arm will also receive a single placebo dose.
  Arm II will receive placebo intraoperatively followed by 3 postoperative doses of thymoglobulin.
  Other Names: thymoglobulin
  Arms: thymoglobulin (postoperative dosing)

SUMMARY:
The purpose of this study is to take a population of lung transplant recipients who meet UCLA criteria for induction chemotherapy with thymoglobulin and prospectively study weather giving the first dose intraoperatively versus postoperatively makes a difference with how patients do during and after lung transplantation.

DETAILED DESCRIPTION:
The purpose of this study is to take a population of lung transplant recipients who meet UCLA criteria for induction chemotherapy with thymoglobulin and prospectively study weather giving the first dose intraoperatively versus postoperatively makes a difference with how patients do during and after lung transplantation. In addition, these cohorts will be compared to patients who do not qualify for thymoglobulin and receive either an alternative agent or no agent. The primary endpoint is primary graft dysfunction. We will also evaluate several other early and late end points such as ventilator days, ICU/hospital days, acute/chronic rejection, infection, CT chest abnormalities, and survival.

We will also collect donor lung tissue and lavage fluid for measurement of various proteins and receptor expression at two time points: (1) prior to implementation and dosing of induction chemotherapy and (2) after transplantation (following a course of induction chemotherapy). This will allow us to possibly make a connection between the profiles of the various proteins and receptors and the clinical outcomes, depending on weather the patient has received induction chemotherapy, starting intraoperatively or postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* On a voluntary basis, all patients eligible for bilateral lung transplantation between the ages of 18-65 years (inclusive)

Exclusion Criteria:

* Have any known allergy to horse or rabbit antithymocyte polyclonal agents
* Have a preoperative platelet count less then 100,000/mm3
* Are recipients of multiple organ transplants (either simultaneous or sequential)
* Are recipients of a single lung transplantation
* Have a contraindication to rabbit antithymocyte globulin based on judgement of the investigators (i.e. bleeding diathesis or overwhelming risk of intense immunosuppression) including the following patients: greater than 65 years of age, prior diagnosis of malignancy (with the exception skin malignancies), underlying suppurative lung disease (i.e. bronchiectasis, cystic fibrosis, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Primary Graft Dysfunction | paO2/FiO2 ratio at post transplant, 24 hr, 48 hr, and 72 hr time points
  the definition for primary graft dysfunction is established and will be used to determine the grade of primary graft dysfunction at 4 time points after lung transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Rajan Saggar, MD, Principal Investigator — Pulmonology & Critical Care at UCLA
Locations (1):
- Departments of Pulmonary and Critical Care, Cardiothoracic Surgery and Infectious Diseases at David Geffen School of Medicine at UCLA, Los Angeles, California, United States